CLINICAL TRIAL: NCT04079062
Title: Single Ascending Dose Study to Assess the Safety, Tolerability, PK and PD of ONO-4685 in Japanese and Caucasian Healthy Adult Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ONO-4685-01
Record Dates: First submitted 2019-08-25; First posted 2019-09-06 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — keyhole-limpet hemocyanin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- ONO-4685 (PartA, D) (Experimental)
  Interventions: Biological: ONO-4685
- Placebo (PartA, D) (Placebo Comparator)
  Interventions: Biological: Placebo
- KLH+placebo (Part B) (Experimental)
  Interventions: Biological: KLH
- KLH+ONO-4685 (PartC) (Experimental)
  Interventions: Biological: KLH, ONO-4685
- KLH+placebo (PartC) (Experimental)
  Interventions: Biological: KLH, placebo

INTERVENTIONS:
Biological: ONO-4685 — Single ascending dose of ONO-4685 will be administered by intravenous continuous infusion at the designated speed.
  Arms: ONO-4685 (PartA, D)
Biological: Placebo — Placebo will be administered by intravenous continuous infusion at the designated speed.
  Arms: Placebo (PartA, D)
Biological: KLH — KLH 1 mg per dose will be subcutaneously administered. In addition, all subjects will be administered placebo after KLH administration.
  Arms: KLH+placebo (Part B)
Biological: KLH, ONO-4685 — Part C will be conducted in a study design that ONO-4685 will be administered within the dose range, for which the safety has been confirmed in Part A, after administering KLH in the dose regimens selected according to the investigation result in Part B.
  Arms: KLH+ONO-4685 (PartC)
Biological: KLH, placebo — Part C will be conducted in a study design that placebo will be administered within the dose range, for which the safety has been confirmed in Part A, after administering KLH in the dose resimens selected according to the investigation result in Part B.
  Arms: KLH+placebo (PartC)

SUMMARY:
To investigate safety, tolerability, pharmacokinetics, pharmacodynamics and immunogenicity in Japanese and Caucasian healthy adult male subjects when ONO-4685 is administered as a single-dose by intravenous infusion.

DETAILED DESCRIPTION:
To investigate safety, tolerability, pharmacokinetics, pharmacodynamics and immunogenicity when ONO-4685 is administered by single-dose intravenous continuous infusion in Japanese and Caucasian healthy adult male subjects. In addition, in Japanese healthy adult male subjects, to investigate dosing condition of Keyhole limpet hemocyanin (KLH) and to investigate safety, tolerability, pharmacokinetics, pharmacodynamics and immunogenicity when ONO-4685 is administered by single-dose intravenous continuous infusion after treating with KLH.

ELIGIBILITY:
Inclusion Criteria:

* Japanese healthy adult male subjects (PartA, B, and C)
* Caucasian healthy adult male subjects (Part D)
* Age (at the time of informed consent): ≥20 yeas, ≤ 45 yeas
* Body weight (at the time of screening test): ≥50 kg

Exclusion Criteria:

* Subjects who are on a treatment for or with a history of respiratory, cardiovascular, psychiatric, neurologic, gastrointestinal, immunologic, hepatic, renal, hematopoietic or endocrine and/or other disease.
* Subjects with current or with a history of severe allergy to drugs or foods
* Subjects with current or with a history of drug or alcohol abuse

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Adverse events [Safety and Tolerability] | Up to 84 days
  Number of participants with adverse events as assessed by CTCAE v5.0
Vital sign [Safety and Tolerability] | Up to 84 days
  Summary statistics of blood pressure/pulse rate, respiratory rate, SpO2
Body temperature [Safety and Tolerability] | Up to 84 days
  Summary statistics of body temperature
Body weight [Safety and Tolerability] | Up to 84 days
  Summary statistics of body weight
ECG parameter test [Safety and Tolerability] | Up to 84 days
  Summary statistics of ECG parameter test (Heart Rate, RR, PR, QRS, QT, and QTcF)
Laboratory test [Safety and Tolerability] | Up to 84 days
  Summary statistics of laboratory test (hematologic test, blood biochemistry test, blood coagulation test, immunoserologic test urinalysis)

SECONDARY OUTCOMES:
Cmax [Pharmacokinetic] (PartA, C, and D) | Up to 84 days
  Assessment of the Cmax of ONO-4685
Tmax [Pharmacokinetic] (PartA, C, and D) | Up to 84 days
  Assessment of the Tmax of ONO-4685
AUC [Pharmacokinetic] (PartA, C, and D) | Up to 84 days
  Assessment of the AUC168h, AUClast, and AUCinf of ONO-4685
T1/2 [Pharmacokinetic] (PartA, C, and D) | Up to 84 days
  Assessment of the T1/2 of ONO-4685
CL [Pharmacokinetic] (PartA, C, and D) | Up to 84 days
  Assessment of the CL of ONO-4685
Vss [Pharmacokinetic] (PartA, C, and D) | Up to 84 days
  Assessment of the Vss of ONO-4685
Serum cytokine concentration [Pharmacodynamics] (PartA, C, and D) | Up to 84 days
  Serum cytokine concentration
Hemocyte test [Pharmacodynamics] (PartA, C, and D) | Up to 84 days
  Hemocyte test
Pharmacodynamics (Part B and C) | Up to 84 days
  Anti-KLH antibody
Immunogenicity (PartA, C, and D) | Up to 84 days
  Anti-ONO-4685 antibody

CONTACTS AND LOCATIONS:
Overall Officials: Junichiro Manako, Study Director — Ono Pharmaceutical Co. Ltd
Locations (1):
- Fukuoka Clinical Site, Hakata, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: No